CLINICAL TRIAL: NCT02035904
Title: Levobupivacaine Prolonged Wound Infusion for Postoperative Pain Relief After Breast Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Massimo Allegri, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011-006331-35
Record Dates: First submitted 2014-01-11; First posted 2014-01-14 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Acute Pain; Chronic Pain; Wound Infusion; Mastectomy
MeSH Terms: conditions — Acute Pain; Chronic Pain | interventions — Sodium Chloride; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levobupivacaine (Experimental): Levobupivacaine Patient Controlled Infusion 5 ml 0,25%, lock out 2 hours
  Interventions: Drug: Levobupivacaine PCIA (Patient Controlled Intrawound Analgesia); Drug: Levobupivacaine continuous infusion; Device: intrawound infusion catheter; Drug: morphine; Drug: Patrol
- Saline (Placebo Comparator): patient controlled infusion 5 ml bolus, lock out 2 hours
  Interventions: Drug: saline; Drug: Levobupivacaine continuous infusion; Device: intrawound infusion catheter; Drug: morphine; Drug: Patrol

INTERVENTIONS:
Drug: Levobupivacaine PCIA (Patient Controlled Intrawound Analgesia) — patient controlled infusion from the 2nd day after surgery
  Arms: Levobupivacaine
Drug: saline — patient controlled infusion from the 2nd day after surgery
  Arms: Saline
Drug: Levobupivacaine continuous infusion — Continuous infusion Levobupivacaine 0,25% 5ml/h for 24 hs in all patients
Device: intrawound infusion catheter — placed by surgeon at the end surgery in all patients
Drug: morphine — PCA with morphine: 0,5 mg/ml bolus 1 mg lock-out 5 min max 20 mg in 4 hs - for the first 24 hs as rescue analgesia
Drug: Patrol — tramadol-paracetamol 37,5/325 mg oral fix combination-rescue analgesia from 2nd day (after morphine PCA removal)

SUMMARY:
The aim of the study is to evaluate efficacy and safety of long term (14 days) wound infusion with levobupivacaine in patients with breast cancer undergoing mastectomy with immediate breast reconstruction: this is a double blind, randomized, parallel group study. The study moves from the concept that nociceptive stimulus last further than 48 hours after surgical intervention: long term analgesia is necessary to provide a real benefit to the patient and provide central sensitization. Intralesional catheter is placed at the end of surgery. In the first 24 postoperative hours we provide continuous wound infusion with levobupivacaine 0,25% 5ml/h with morphine Patient Controlled Analgesia (PCA) when NRS >4. From the second postoperative day morphine PCA is removed and patients are randomized to receive levobupivacaine 0,25% or saline, released with 5 ml boluses and lock-out of 2 hours, with rescue analgesia with tramadol 37,5 mg + acetaminophen 325 mg oral fix combination (Patrol). Intralesional catheter is taken off 14 days after surgical intervention or after 36 hours of non-use.

Pain evaluation (NRS at rest and movement) and oral rescue doses consumption are performed; pain physicians also care about any catheter-related or drug-related side effect, registering number of total boluses. Patients are provided with a home diary for pain scores to be filled and brought back when surgical visit is performed. A phone interview at 1 and 3 month is performed to investigate pain chronicization.

Surgical evaluation is provided, also to establish any catheter-related infective or healing complication.

Physiatric evaluation before the intervention and 1 and 3 months is provided to ensure rehabilitation process.

A validated questionnaire (short form 36/ SF-36) must be filled by all patients, to understand differences in return to a normal quality of life and to social activities between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* F; age 18 to 70
* American Society of Anesthesiologists (ASA) I e II;
* breast cancer ( DIN 2 e 3, o LIN 2 e 3 sec. Tavassoli) scheduled for nipple-sparing mastectomy, simple mastectomy, skin-sparing mastectomy, skin-reducing mastectomy c, lymphnode biopsy and axillary dissection;
* immediate sub-pectoral prosthetic reconstruction;
* signed informed consent.

Exclusion Criteria:

* preexisting pectoral, axillar, thoracic homolateral pain
* habitual opioid consumption;
* drug-alcoholics addiction ;
* ICU postoperative recovery;
* kidney failure (creatinin > 2 g/dl, creatinin <clearance 30 ml/h) and/or hepatic failure (cholinesterase < 2000 UI);
* cardiac arrhythmias o;
* Epilepsy;
* Psychiatric, cognitive disorders, mental retardation;
* Coagulopathies (INR > 2, activated partial thromboplastin time - aPTT>44 sec);
* platelet count less than 100.000/mm3;
* BMI > 30;
* Allergies to study drugs.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
reduction in oral Tramadol-Paracetamol combination consumption from 2nd to 14th day after mastectomy | from day 2 to 14

SECONDARY OUTCOMES:
reduction in pain values at rest and movement in treatment group | 14 days
incidence of drug-related side effects | up to 14 days
  local anesthetic toxicity, opioid side effects
incidence of catheter-related surgical complications | up to 1 month
  infections, healing retardation
earlier upper limb rehabilitation | up to 1 month
  physiatric evaluations
earlier return to social activities and good quality of life | up to 1 month
  validated SF-36 questionnaire
different chronic pain incidence | up to 3 months
  phone interview at 1 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Allegri Massimo, MD, Principal Investigator — Pain Therapy Service IRCCS Policlinico S Matteo Pavia Italy
Locations (1):
- Department of Anesthesia - Pain Therapy Service, Pavia, Pavia, Italy